CLINICAL TRIAL: NCT03183128
Title: A Phase 3 Multicenter, RandomizeEd, Double Blind, Placebo COntrolled, Parallel Group Study to Evaluate the Safety, Tolerability, & Efficacy of SER-109 vs. Placebo to Reduce Recurrence of ClOstRidium Difficile Infection (CDI) in Adults
Brief Title: ECOSPOR III - SER-109 Versus Placebo in the Treatment of Adults With Recurrent Clostridium Difficile Infection
Acronym: ECOSPORIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seres Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERES-012
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2021-06

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SER-109 (Experimental): Received oral dose of SER-109
  Interventions: Biological: SER-109
- Placebo (Placebo Comparator): Received matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: SER-109 — SER-109 is an ecology of bacteria in spore form, enriched from stool donations obtained from healthy, screened donors
  Other Names:
  Eubacterial Spores, Purified Suspension, Encapsulated
  Arms: SER-109
Drug: Placebo — Placebo will be identical to the investigational product but will not contain product spores or non-spore solids. Placebo will consist of 92% glycerol and 8% normal saline(0.9%).
  Arms: Placebo

SUMMARY:
Subjects will receive an oral dose of SER-109 in 4 capsules once daily for 3 consecutive days in Treatment Group I or matching placebo once daily for 3 consecutive days in Treatment Group II. The purpose of this study is to demonstrate the superiority of SER-109 vs placebo to reduce recurrence of CDI as determined by a toxin assay in adults up to 8 weeks after initiation of treatment.

DETAILED DESCRIPTION:
ECOSPOR III is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study of the safety, tolerability, and efficacy of SER-109 versus placebo in adult subjects 18 years of age or older with recurrent CDI, defined as: a history of ≥ 3 CDI episodes within 12 months, inclusive of the current episode. This study is designed to demonstrate the superiority of SER-109 versus placebo to reduce recurrence of Clostridium difficile infection (CDI) in adults who have received antibacterial drug treatment for recurrent CDI (RCDI), based on the proportion of subjects experiencing a CDI recurrence requiring antibiotic treatment up to 8 weeks after initiation of treatment. Approximately 188 subjects with a history of CDI, diarrhea and a positive C. difficile toxin test result on a stool sample, who have responded to standard-of-care (SOC) antibiotic treatment will be enrolled. Subjects will be randomly assigned, in a 1:1 ratio, to 1 of 2 treatment groups (Treatment Group I [SER-109] or Treatment Group II [Placebo]) and stratified by age (<65 years; ≥65 years), as well as antibiotic regimen for the qualifying episode (vancomycin; fidaxomicin).

Subjects will receive an oral dose of SER-109 in 4 capsules once daily for 3 consecutive days in Treatment Group I or matching placebo once daily for 3 consecutive days in Treatment Group II.

Subjects with confirmed CDI recurrence, as defined in the Protocol, up to 8 weeks after administration of SER-109 or placebo treatment, may be eligible to enroll in the open-label SER-109 extension study (Study SERES-013).

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-specific procedure or treatment. The subject or their legally authorized representative must be able to provide written informed consent and understand the potential risks and benefits from study enrollment and treatment.
2. Male or female subject ≥ 18 years of age.
3. A qualifying episode of CDI as defined by:

   1. ≥ 3 unformed stools per day for 2 consecutive days
   2. A positive C. difficile stool toxin assay.
   3. The requirement of CDI SOC antibiotic therapy (defined as 10 to 21 days of treatment with vancomycin [125 mg QID] and/or fidaxomicin [200 mg BID]).
   4. An adequate clinical response following SOC antibiotic therapy, defined as (<3 unformed stools in 24 hours) for 2 or more consecutive days before randomization.

Main Exclusion Criteria:

1. Female subjects who are pregnant, breastfeeding, lactating, or planning to become pregnant during the study.
2. Known or suspected toxic megacolon and/or known small bowel ileus.
3. Admitted to or expected to be admitted to an intensive care unit for medical reasons (not just boarding). Note: nursing homes, rehabilitation, assisted living centers and acute care hospitals are acceptable.
4. Absolute neutrophil count of <500 cells/ml^3
5. Major gastrointestinal surgery (e.g. significant bowel resection or diversion) within 3 months before enrollment (this does not include appendectomy or cholecystectomy), or any history of total colectomy or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, i.e., restrictive procedures such as banding, are permitted).
6. History of active inflammatory bowel disease (ulcerative colitis, Crohn's disease, microscopic colitis) with diarrhea believed to be caused by active inflammatory bowel disease in the past 3 months.
7. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy (subjects on maintenance chemotherapy may only be enrolled after consultation with the study medical monitor).
8. Any history of fecal microbiota transplantation (FMT) within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa von Moltke, MD, Study Director — Seres Therapeutics, Inc.
Locations (54):
- United States (49):
  - (Investigator site), North Little Rock, Arkansas
  - (Investigator site), Mather, California
  - (Investigator site), Mountain View, California
  - (Investigator site), Northridge, California
  - (Investigator site), Sacramento, California
  - (Investigator site), Simi Valley, California
  - (Investigator site), Upland, California
  - (Investigator site), Hamden, Connecticut
  - (Investigator site), Washington D.C., District of Columbia
  - (Investigator site), Jacksonville, Florida
  - (Investigator site), Miami, Florida
  - (Investigator site), Pembroke Pines, Florida
  - (Investigator site), Athens, Georgia
  - (Investigator site), Atlanta, Georgia
  - (Investigator site), Marietta, Georgia
  - (Investigator site), Riverdale, Georgia
  - (Investigator site), Sandy Springs, Georgia
  - (Investigator site), Idaho Falls, Idaho
  - (Investigator site), Springfield, Illinois
  - (Investigator site), Evansville, Indiana
  - (Investigator site), Jeffersonville, Indiana
  - (Investigator site), Iowa City, Iowa
  - (Investigator site), Kansas City, Kansas
  - (Investigator site), New Orleans, Louisiana
  - (Investigator site), Annapolis, Maryland
  - (Investigator site), Chevy Chase, Maryland
  - (Investigator site), Boston, Massachusetts
  - (Investigator site), Worcester, Massachusetts
  - (Investigator site), Detroit, Michigan
  - (Investigator site), Royal Oak, Michigan
  - (Investigator site), St Louis, Missouri
  - (Investigator site), Butte, Montana
  - (Investigator site), Las Vegas, Nevada
  - (Investigator site), Buffalo, New York
  - (Investigator site), Greenville, North Carolina
  - (Investigator site), Kinston, North Carolina
  - (Investigator site), Raleigh, North Carolina
  - (Investigator site), Centerville, Ohio
  - (Investigator site), Cleveland, Ohio
  - (Investigator site), Columbus, Ohio
  - (Investigator site), Pittsburgh, Pennsylvania
  - (Investigator site), Sayre, Pennsylvania
  - (Investigator site), Houston, Texas
  - (Investigator site), San Antonio, Texas
  - (Investigator site), Southlake, Texas
  - (Investigator site), Bountiful, Utah
  - (Investigator site), Riverton, Utah
  - (Investigator site), Charlottesville, Virginia
  - (Investigator site), Reston, Virginia
- Canada (5):
  - (Investigator site), Calgary, Alberta
  - (Investigator site), Vancouver, British Columbia
  - (Investigator site), Victoria, British Columbia
  - (Investigator site), London, Ontario
  - (Investigator site), Chicoutimi, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bryant JA, Vulic M, Walsh EA, Allen EG Jr, Beauchemin NJ, Chafee ME, Diao L, Fenn K, Ford KA, Hasson BR, Litcofsky KD, Lombardo MJ, Martinez A, O'Brien EJ, Straub TJ, Sykes SM, Marshall LF, Winkler JA, McGovern BH, Ford CB, Wortman JR, Henn MR. The impact of an oral purified microbiome therapeutic on the gastrointestinal microbiome. Nat Med. 2026 Jan;32(1):186-196. doi: 10.1038/s41591-025-04076-w. Epub 2026 Jan 5. PMID 41491103
- [Derived] Kraft CS, Sims M, Silverman M, Louie TJ, Feuerstadt P, Huang ES, Khanna S, Berenson CS, Wang EEL, Cohen SH, Korman L, Lee C, Kelly CR, Odio A, Cook PP, Lashner B, Ramesh M, Kumar P, De A, Memisoglu A, Lombardi DA, Hasson BR, McGovern BH, von Moltke L, Pardi DS; ECOSPOR III and ECOSPOR IV investigators. Integrated Safety and Efficacy Analyses of Phase 3 Trials of a Microbiome Therapeutic for Recurrent CDI. Infect Dis Ther. 2024 Oct;13(10):2105-2121. doi: 10.1007/s40121-024-01007-z. Epub 2024 Jun 28. PMID 38941068
- [Derived] Garey KW, Jo J, Gonzales-Luna AJ, Lapin B, Deshpande A, Wang E, Hasson B, Pham SV, Huang SP, Reese PR, Wu H, Hohmann E, Feuerstadt P, Oneto C, Berenson CS, Lee C, McGovern B, vonMoltke L. Assessment of Quality of Life Among Patients With Recurrent Clostridioides difficile Infection Treated with Investigational Oral Microbiome Therapeutic SER-109: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2253570. doi: 10.1001/jamanetworkopen.2022.53570. PMID 36716031
- [Derived] Feuerstadt P, Louie TJ, Lashner B, Wang EEL, Diao L, Bryant JA, Sims M, Kraft CS, Cohen SH, Berenson CS, Korman LY, Ford CB, Litcofsky KD, Lombardo MJ, Wortman JR, Wu H, Aunins JG, McChalicher CWJ, Winkler JA, McGovern BH, Trucksis M, Henn MR, von Moltke L. SER-109, an Oral Microbiome Therapy for Recurrent Clostridioides difficile Infection. N Engl J Med. 2022 Jan 20;386(3):220-229. doi: 10.1056/NEJMoa2106516. PMID 35045228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, there were 51 sites in the United States and 5 sites in Canada that enrolled participants between 2017 to 2020.
Groups:
- SER-109: Randomized to SER-109 arm. Assigned to receive SER-109 oral dose of 4 capsules once daily for 3 consecutive days.
- Placebo: Randomized to matching Placebo arm. Assigned to receive Placebo oral dose of 4 capsules once daily for 3 consecutive days.
Period: Overall Study
Arm/Group | SER-109 | Placebo
Started ("Started" represents the number of participants assigned to each arm. Note: The number of participants who actually received SER-109 was 90, and those who actually received Placebo was 92.) | 89 | 93
Completed 8-Week Follow-up | 84 | 65
Completed (Completed 24-Week Follow-up) | 77 | 56
Not Completed | 12 | 37
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Protocol Violation | 2 | 0
Not completed — Lack of Efficacy | 4 | 27
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SER-109 | Placebo | Total
Number analyzed (Participants) | 89 | 93 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (16.5) | 65.5 (16.7) | 65.5 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 49 | 109
  Male | 29 | 44 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 82 | 88 | 170
  Other | 2 | 1 | 3
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 84 | 87 | 171
Antibiotic regimen for qualifying episode [Count of Participants; unit: Participants]
  Vancomycin | 64 | 69 | 133
  Fidaxomicin | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of CDI up to 8 Weeks
Description: Recurrence of CDI up to 8 Weeks after initiation of treatment. Recurrence was determined by stool Clostridioides difficile toxin assay.
Time Frame: Up to Week 8
Population: All participants who were randomly assigned, including those who were not exposed to any study drug, were analyzed based on the treatment to which they were randomly assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 89 | 93
Participants | 11 | 37
Statistical Analysis 1: Comparison: SER-109 vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value presented for both hypothesis tests: H0: RR≥1 and H0: RR≥0.833; Cochran-Mantel-Haenszel test was stratified by age (<65 years, ≥65 years) and prior antibiotic regimen (vancomycin, fidaxomicin); Risk Ratio (RR) = 0.32, 95% CI 2-sided [0.18 to 0.58] — RR defined as the recurrence rates of SER-109 divided by Placebo. Cochran-Mantel-Haenszel estimate of RR, stratified by age group (<65 years, ≥65 years) and prior antibiotic regimen for the qualifying episode (vancomycin, fidaxomicin), is reported

2. Secondary Outcome: Recurrence of CDI up to 4, 12 and 24 Weeks
Description: Recurrence of CDI up to 4, 12 and 24 Weeks after initiation of treatment. Recurrence was determined by stool Clostridioides difficile toxin assay.
Time Frame: Up to 4, 12 and 24 weeks after treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 89 | 93
Participants
  CDI Recurrence-Week 4 | 10 | 31
  CDI Recurrence-Week 12 | 16 | 43
  CDI Recurrence-Week 24 | 19 | 44
Statistical Analysis 1: Comparison: SER-109 vs Placebo; CDI recurrence rates at Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value presented is for the hypothesis test: H0: RR ≥1.0; The Cochran-Mantel-Haenszel estimate is stratified by age (<65 years, ≥65 years) and prior antibiotic regimen (vancomycin, fidaxomicin); Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.19 to 0.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: SER-109 vs Placebo; CDI recurrence rates at Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value presented is for the hypothesis test: H0: RR ≥1.0; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.24 to 0.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: SER-109 vs Placebo; CDI recurrence rates at Week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value presented is for the hypothesis test: H0: RR ≥1.0; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.30 to 0.73] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 24-week follow-up
Description: Participants were analyzed according to the treatment they actually received. Two subjects were originally assigned to SER-109 arm, but received Placebo, while 3 subjects were originally assigned to Placebo arm, but received SER-109.
  All adverse events were collected from Day 1 post-dosing to Week 8. From Week 8 to the end of study (Week 24), only serious adverse events and adverse events of special interest (i.e., invasive infections) were collected.
Groups:
- SER-109: Received SER-109 oral dose of 4 capsules once daily for 3 consecutive days
- Placebo: Received matching Placebo oral dose of 4 capsules once daily for 3 consecutive days
Arm/Group | SER-109 | Placebo
All-Cause Mortality (participants affected / at risk) | 3/90 | 0/92
Serious Adverse Events (participants affected / at risk) | 15/90 | 19/92
Other Adverse Events (participants affected / at risk) | 77/90 | 79/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SER-109 (N=90) | Placebo (N=92)
Urinary tract infection (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Clostridioides difficile colitis (Infections and infestations) | 1 | 7
Cystitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Bacterial colitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Sclerites (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SER-109 (N=90) | Placebo (N=92)
Abdominal distension (Gastrointestinal disorders) | 49 | 49
Abdominal pain (Gastrointestinal disorders) | 46 | 56
Constipation (Gastrointestinal disorders) | 28 | 22
Diarrhea (Gastrointestinal disorders) | 22 | 20
Flatulence (Gastrointestinal disorders) | 63 | 70
Nausea (Gastrointestinal disorders) | 16 | 30
Chills (General disorders) | 21 | 22
Fatigue (General disorders) | 53 | 58
Urinary tract infection (Infections and infestations) | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 26 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03183128/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03183128/SAP_001.pdf